CLINICAL TRIAL: NCT06381882
Title: Establishing the Role of the Human Microbiome in Patients With a Presumed Pancreatic or Periampullary (Pre)Malignancy and Pancreatic Resection.
Brief Title: The Role of the Human Microbiome in Patients After Pancreatic Resection.
Acronym: MiPac
Status: Not yet recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Robert Verdonk, dr., St. Antonius Hospital
Other Study IDs: MiPac
Record Dates: First submitted 2024-02-25; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm; Pancreas Adenocarcinoma; Periampullary Cancer; Periampullary Carcinoma; Microbial Colonization
MeSH Terms: conditions — Pancreatic Neoplasms; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Faeces
  * Rectal swab
  * Blood (full)
  * Tumor
  * Saliva
  * Bile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Adult patients with resectable pancreatic or periampullary presumed (pre)malignancy
  Interventions: Procedure: Pancreatic resection

INTERVENTIONS:
Procedure: Pancreatic resection — Any kind of pancreatic resection will be included

SUMMARY:
The goal of this observational study is to classify patients that undergo pancreatic resection for presumed pancreatic or periampullary malignancy into high and low risk groups for postoperative complications based on longitudinal saliva, rectal/faecal, tumor, blood and/or bile microbiome profiles.

To identify the dynamics of the microbiome, as well as the possibly related short-term and long-term complications, multiple samples at different timepoints are needed from the patients.

DETAILED DESCRIPTION:
Rationale:

Resection is the only potentially curative option for pancreatic and periampullary cancer, a complex procedure with a high risk of complications of 30% to 73%. Research shows the presence of altered bacterial populations within fecal, pancreatic fluid, bile and jejunal samples of patients after pancreatic resection compared to healthy samples. Moreover, specific gut microbial composition in the pre- and postoperative period were associated with a higher risk of developing complications after pancreatic resection in small studies. Further research on a larger scale is necessary to validate these findings and to evaluate targeted microbiome modifications to improve outcomes in patients after pancreatic resection.

Objective:

The primary objective of this study is to classify patients that undergo pancreatic resection for presumed pancreatic or periampullary malignancy into high and low risk groups for postoperative complications based on longitudinal microbiome profiles.

Study design: Prospective observational cohort study.

Study population: 200 adult patients with resectable pancreatic or periampullary presumed (pre)malignancy.

Main study parameters/endpoints:

The primary endpoint is a composite of postoperative complications including pancreatic fistula, bleeding, gastroenterostomy-, bile- or chyle leakage, delayed gastric emptying, cholangitis, sepsis and organ failure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

All participants will be offered the standard of care. In addition, rectal swabs, faeces, salivary, bile, blood and tumor samples will be collected at different time points perioperatively. Participating in this study carries no additional risks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with a resectable, borderline resectable or locally advanced pancreatic and periampullary presumed (pre)malignancy.
* The intention of the treatment must be curative including surgery and (neo-)adjuvant chemotherapy.
* Willing and able to adhere to the study procedures described in this protocol and to grant the study team access to the electronic patient file and other data that are required to answer the research questions described in this protocol.

Exclusion Criteria:

* Inability to provide adequate informed consent (e.g. language barrier, illiteracy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises of adult patients that are presented at the Regional Academic Cancer Center Utrecht (RAKU) with a pancreatic or periampullary presumed (pre)malignancy, where diagnosis must be established at the regional multidisciplinary meeting and the intention of the treatment must be curative.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Risk stratification postoperative complications | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  The primary objective of this study is to classify patients that undergo pancreatic resection into high and low risk groups for postoperative complications, based on saliva, blood, tumor, bile and/or rectal/faecal microbiome profiles.

SECONDARY OUTCOMES:
Long time oncological outcomes - site of recurrence | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and long term oncological outcomes (e.g. site of recurrence).
Long time oncological outcomes - disease free survival | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and long term oncological outcomes (e.g. disease free survival).
Long time oncological outcomes - overall survival | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and long term oncological outcomes (e.g. overall survival).
Complications neoadjuvant chemotherapy | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and complications of neoadjuvant chemotherapy.
Complications adjuvant chemotherapy | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and complications of adjuvant chemotherapy.
Response to neoadjuvant chemotherapy | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and response to neoadjuvant chemotherapy as judged by computed tomography (CT) scan and histological respons.
Complications bile duct drainage | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and complications associated with bile duct drainage.
Postoperative endocrine insufficiency | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and postoperative endocrine insufficiency (defined as need for new pharmacologic intervention).
Postoperative exocrine insufficiency | - (Before start chemotherapy), peroperative, preoperative, postoperative day 1/3, +/- 2 weeks post-discharge
  Secondary objectives include, but are not limited to, finding associations between microbiome profiles and postoperative exocrine insufficiency (defined as need for new pharmacologic intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Verdonk, dr., Principal Investigator — St. Antonius Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan is to be discussed.